CLINICAL TRIAL: NCT04940247
Title: Myocardial Perfusion Imaging by Combined 15O-H2O PET and MR for Evaluation of Reversible Myocardial Ischemia
Brief Title: Myocardial Perfusion Imaging by Combined 15O-H2O PET and MR
Acronym: PREFER
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PREFER
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Heart Disease
Keywords: Myocardial perfusion imaging; Positron-Emission Tomography; Cardiac Magnetic Resonance Imaging; Coronary Artery Disease; Coronary Flow Reserve; Myocardial Blood Flow
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial will include 75 patients with evident or suspected ischemic heart disease refered to Department of Nuclear Medicine & PET Centre, Aarhus University Hospital, for perfusion imaging by 15O-H2O PET/CT scan of the heart during rest and stress. Instead of the clinical scan participants will undergo perfusion imaging by 15O-H2O PET/MR.

The clinician will receive diagnostic information based on the 15O-H2O PET scan as if the patient had not participated in the study. As such, the study has no influence on the diagnostics or treatments of the patient.

Data from the scans will be used to compare 15O-H2O PET with cardiac MR for evaluation of myocardial perfusion.

Follow up will be done for up to 10 years in regards to major cardiovascular events in order to determine the prognostic value of the scan.

ELIGIBILITY:
Inclusion Criteria:

* Refered for myocardial perfusion imaging by O15-H2O PET at Department of Nuclear Medicine & PET Centre, Aarhus University Hospital
* > 18 years of age

Exclusion Criteria:

* Allergic to adenosine
* Allergic to gadolinium
* Pregnancy
* Claustrophobia
* Severe Asthma
* Pacemaker or other ferro-magnetic implants
* GFR < 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with known or suspected ischemic heart disease referred for a clinical H2O-PET at Department of Nuclear Medicine and PET Centre, Aarhus University Hospital, not meeting any exclusion criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Difference in myocardial blood flow | 2 years
  The difference in assessed myocardial blood flow as measured by 15O-H2O PET and MR
Prognostic value within 10 years | 10 years
  Number of participants who experience a major adverse cardiac event within 10 years of follow-up.

SECONDARY OUTCOMES:
Difference in coronary flow reserve | 2 Years
  The difference in assessed myocardial blood flow as measured by 15O-H2O PET and MR
Difference in predictive value | 10 years
  The difference in predictive value of myocardial blood flow measurements as measured by 15O-H2O PET and MR
Difference in left ventricular end-systolic volume | 2 years
  The difference in left ventricular end-systolic volume as measured by 15O-H2O PET and MR
Difference in left ventricular end-diastolic volume | 2 years
  The difference in left ventricular end-diastolic volume as measured by 15O-H2O PET and MR
Difference in right ventricular end-systolic volume | 2 years
  The difference in right ventricular end-systolic volume as measured by 15O-H2O PET and MR
Difference in right ventricular end-diastolic volume | 2 years
  The difference in right ventricular end-diastolic volume as measured by 15O-H2O PET and MR
Difference in left ventricular mass | 2 years
  The difference in left ventricular mass as measured by 15O-H2O PET and MR
Amount of scar tissue | 2 years
  Scar tissue assessment as measured by MR
Pulmonary transit time | 2 years
  Pulmonary transit time as measured by 15O-H2O PET
Pulmonary perfusion | 2 years
  Pulmonary perfusion as measured by 15O-H2O PET
Prognostic value within 3,5 years | 5 years
  Number of participants who experience a major adverse cardiac event within 3,5 years of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus N, Denmark